CLINICAL TRIAL: NCT01541579
Title: A Phase III, Randomized, Double Blind, Parallel Group, Placebo Controlled, Multicentre Study to Assess Efficacy and Safety of Expanded Allogeneic Adipose-derived Stem Cells (eASCs) for the Treatment of Perianal Fistulising Crohn's Disease Over a Period of 24 Weeks and an Extended Follow-up Period up to 104 Weeks.
Brief Title: Adipose Derived Mesenchymal Stem Cells for Induction of Remission in Perianal Fistulizing Crohn's Disease
Acronym: ADMIRE-CD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cx601-0302
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Crohn's Disease
Keywords: Perianal fistulising Crohn's disease.
MeSH Terms: conditions — Crohn Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Cx601 is a cell suspension in aseptic buffered solution containing human expanded adipose-derived stem cells (eASCs) of allogeneic origin in disposable vials with no preservative agents. The cells will be given at a dose of 120 million cells (5 million cells / mL) for intralesional injection.
  Interventions: Other: Cx601
- Placebo-control group (Placebo Comparator): Placebo (saline solution) will be given also for intralesional injection at the same quantity (volume, 24 mL) and following the same schedule.
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Cx601 — 120 million cells administered by intralesional injection.
  Arms: Treatment Arm
Other: Saline solution — 24 mL saline solution by intralesional injection
  Arms: Placebo-control group

SUMMARY:
The current multicentre phase III study is proposed to confirm in an add-on therapy design compared to a placebo-control group, the efficacy of adipose-derived stem cells (eASCs) from healthy donors for the treatment of complex anal fistulas in patients with Crohn's disease over a 24-week period and an extended follow-up period up to 104 weeks.

DETAILED DESCRIPTION:
The current multicentre phase III study is proposed to confirm in an add-on therapy design compared to a placebo-control group, the efficacy of adipose-derived stem cells (eASCs) from healthy donors for the treatment of complex anal fistulas in patients with Crohn's disease over a 24-week period and an extended follow-up period up to 104 weeks. Subject with perianal fistulising Crohn's disease will be treated with Cx601, suspension of eASCs, at a dose of 120 million cells administered by intralesional injection. The treatment of complex perianal fistulas by local application of eASCs intends to improve significantly the local conditions with very few inconveniences (ambulatory procedure) and minimal risk of possible complications (anal incontinence). Therefore, this is a new therapeutic resource that is expected to be safe and efficacious as well as is expected to improve the quality of life of the patients in this highly debilitating and chronic condition. This treatment would prevent one of the main causes of anal incontinence, would diminish recurrence of the fistula disease and would reduce drastically the significant disorders provoked by the standard fistula surgery in the patients. Indeed, patients can be discharged according to the "One Day Surgical" procedures (major ambulatory surgery).

ELIGIBILITY:
Inclusion Criteria:

The reference population will consist of patients with perianal fistulising Crohn´s disease refractory to at least one of the following treatments: antibiotics, immunosuppressants or anti-tumor necrosis factor (TNF). Naïve patients are excluded, and those patients refractory to antibiotics will represent less than 25% of the total recruited patients.

All of them must comply with the following inclusion criteria:

1. Signed informed consent.
2. Patients with Crohn's Disease (CD) diagnosed at least 6 months earlier in accordance with accepted clinical, endoscopic, histological and/or radiologic criteria.
3. Presence of complex perianal fistulas with a maximum of 2 fistulas (internal openings) and a maximum of 3 external openings, assessed by clinical assessment and MRI. Fistula must have been draining for at least 6 weeks prior to the inclusion. A complex perianal fistula is defined as a fistula that met one or more of the following criteria during its evolution:

   * High inter-sphincteric, trans-sphincteric, extra-sphincteric or supra-sphincteric.
   * Presence of ≥ 2 external openings (tracts).
   * Associated collections
4. Non-active or mildly active luminal CD defined by a CDAI ≤ 220.
5. Patients of either sex aged 18 years or older
6. Good general state of health according to clinical history and a physical examination.
7. For women of a childbearing age, they must have negative serum or urine pregnancy test (sensitive to 25 IU human chorionic gonadotropin (hCG)). Both men and women should use appropriate birth control methods defined by the investigator.

Exclusion Criteria:

1. Presence of dominant luminal active Crohn's disease requiring immediate therapy.
2. CDAI >220.
3. Concomitant rectovaginal fistulas
4. Patient naïve to specific treatment for perianal fistulising Crohn's disease including antibiotics
5. Presence of an abscess or collections > 2 cm, unless resolved in the preparation procedure (week -3 to day 0).
6. Presence of > 2 fistular lesions.
7. Presence of > 3 external openings.
8. Rectal and/or anal stenosis and / or active proctitis, if this means a limitation for any surgical procedure.
9. Patient who underwent surgery for the fistula other than drainage or seton placement.
10. Patient with diverting stomas
11. Patient with ongoing steroid treatment or treated with steroids in the last 4 weeks
12. Renal impairment defined by creatinine clearance below 60 ml/min calculated using Cockcroft-Gault formula or by serum creatinine ≥ 1.5 x upper limit of normality (ULN)
13. Hepatic impairment defined by both of the following laboratory ranges:

    * Total bilirubin ≥ 1.5 x ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase(ALT) ≥ 2.5 x ULN
14. Known history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion.
15. Malignant tumour or patients with a prior history of any malignant tumour, including any type of fistula carcinoma.
16. Current or recent history of abnormal, severe, progressive, uncontrolled hepatic, haematological, gastrointestinal (except CD), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral disease.
17. Congenital or acquired immunodeficiencies.
18. Known allergies or hypersensitivity to antibiotics including but not limited to penicillin, streptomycin, gentamicin, aminoglycosides; Human Serum Albumin (HSA); Dulbecco Modified Eagle's Medium (DMEM); materials of bovine origin; local anaesthetics or gadolinium (MRI contrast).
19. Contraindication to MRI scan, (e.g., due to the presence of pacemakers, hip replacements or severe claustrophobia).
20. Major surgery or severe trauma within the previous 6 months.
21. Pregnant or breastfeeding women.
22. Patients who do not wish to or cannot comply with study procedures.
23. Patients currently receiving, or having received within 3 months prior to enrolment into this clinical study, any investigational drug.
24. Patients previously treated with eASCs can not be enrol into this clinical study.
25. Subjects who need surgery in the perianal region for reasons other than fistulas at the time of inclusion in the study, or for whom such surgery is foreseen in this region in the 24 weeks after treatment administration.
26. Contraindication to the anaesthetic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Combine remission of perianal fistulising Crohn's | 24 weeks
  Combined Remission of perianal fistulising Crohn's disease defined as the clinical assessment of closure of all treated external openings (EO) that were draining at baseline despite gentle finger compression at week 24, and absence of collections > 2 cm of the treated perianal fistulas confirmed by centrally blinded MRI assessment by week 24.

SECONDARY OUTCOMES:
Efficacy Assessment by week 24 | 24 weeks
  * Clinical Remission (CR) defined as closure of all treated EO that were draining at baseline despite gentle finger compression, as clinically assessed
  * Response defined as closure of at least 50% of all treated EO that were draining at baseline, as clinically assessed
  * Time to Clinical Remission (time from treatment start to 1st visit with closure of all treated EO as described above)
  * Time to Response (time from treatment start to 1st visit with closure of at least 50% of all treated EO as described above)
  * Relapse defined, in patients with CR at previous visit, as reopening of any of the treated EO with active drainage, or the development of a perianal collection > 2 cm of the treated perianal fistulas confirmed by centrally blinded MRI
  * Time to Relapse in patients with CR (time from CR to 1st visit with reopening of any of the treated EO as described above)
  * Severity of the perianal CD, assessed with the PDAI
  * QoL assessed by IBDQ
  * CDAI score
  * Van Assche
Efficacy Assessment by week 52 | 52 weeks
  * Combined Remission of perianal fistulising Crohn's disease at week 52 (as defined for week 24)
  * Clinical Remission defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression, as clinically assessed at week 52
  * Response defined as closure of at least 50% of all treated external openings that were draining at baseline, as clinically assessed at week 52
  * Time to Combined Remission by week 52 (as defined for week 24)
  * Time to Clinical Remission by week 52 (as defined for week 24)
  * Time to Response by week 52 (as defined for week 24)
  * Relapse by week 52 in patients with Combined Remission at week 24 (as defined for week 24)
  * Time to Relapse by week 52 in patients with Combined Remission at week 24 (as defined for week 24)
  * Severity of the perianal Crohn's disease up to week 52 assessed PDAI
  * QoL up to week 52 by the IBDQ
  * CDAI score up to week 52
  * Van Assche score up to week 52
Efficacy Assessment by week 104 | 104 Weeks
  * Clinical Remission of perianal fistulising Crohn's disease defined as the clinical assessment of closure of all treated external openings that were draining at baseline despite gentle finger compression at week 104
  * Relapse by week 104 in patients with Combined Remission at week 52, defined as reopening of any of the treated external openings with active drainage as clinically assessed
  * Time to Relapse by week 104 in patients with Combined Remission at week 52 (defined as time from Combined Remission to first visit with reopening of any of the treated external openings with active drainage as clinically assessed)
  * Severity of the perianal Crohn's disease, assessed with the Perianal Disease Activity Index (PDAI) up to week 104
  * Quality of Life (QoL) assessed by the Inflammatory Bowel Disease Questionnaire (IBDQ) up to week 104
  * CDAI score up to week 104
Safety analysis throughout the study: | week 24, 52 and 104
  * Adverse events including: Treatment emergent Adverse Events (TEAEs), TEAEs related to study treatment, Treatment emergent Serious Adverse Events (TESAEs), TESAEs related to study treatment, TEAEs leading to study withdrawal, adverse events related to surgical procedure(s) to provide study treatment, deaths Only SAEs will be reported during the 2nd follow-up period between week 52 and week 104.
  * Physical examination
  * Vital signs
  * Laboratory tests (biochemistry, haematology, urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Panes, MD, Study Chair — Hospital Clinic of Barcelona; Julian Panes, MD, Principal Investigator — Hospital Clinic of Barcelona; Lili Kazemi-Shirazi, Professor, Principal Investigator — Medical University of Vienna; Karl Mrak, MD, Principal Investigator — Krankenhaus, St. Veit/Glan; Marc Ferrante, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Kurt Van der Speeten, MD, Principal Investigator — Hospital Oost-Limburg, Genk; Danny de Looze, Professor, Principal Investigator — Gent University Hospital; Filip Baert, MD, Principal Investigator — Hospital Hartziekenhuis, Roeselare; Daniel C Baumgart, Professor, Principal Investigator — Charite University, Berlin, Germany; Axel Dignass, Professor, Principal Investigator — Kilikum Frankfurt; Max Reinshagen, Professor, Principal Investigator — Kinikum Braunschweig; Silvio Danese, MD, Principal Investigator — Instituto Clinico Humanitas IRCCS, Milano; Vito Annese, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi; Anna Kohn, MD, Principal Investigator — Azienda Ospedaliera San Camillo-Forlanini, Rome; Alfredo Papa, MD, Principal Investigator — Università Cattolica del Sacro Cuore, Rome; Giacomo C Sturniolo, Professor, Principal Investigator — Azienda Ospedaliera di Padova; Andrea Belluzi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant'Orsola Malpighi; Gabriele Riegler, Professor, Principal Investigator — University of Campania Luigi Vanvitelli; Bas Oldenburg, MD, Principal Investigator — UMCU, Utrecht; Adriaan A van Bodegraven, MD, Principal Investigator — Amsterdam UMC, location VUmc; Gigs van den Brink, Professor, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); María D Martín Arranz, MD, Principal Investigator — Hospital Universitario La Paz; Jose M Gallardo Valverde, MD, Principal Investigator — Hospital Universitario Reina Sofía, Cordoba; Javier Pérez Gisbert, MD, Principal Investigator — Hospital La Princesa, Madrid; Belén Beltrán Niclós, MD, Principal Investigator — Hospital Universitario La Fe; Carlos Taxonera Samsó, MD, Principal Investigator — Hospital Clínico San Carlos, Madrid; Fernando de la Portilla de Juan, MD, Principal Investigator — Hospital Virgen del Rocío, Seville; Ricardo Rada Morgades, MD, Principal Investigator — Hospital Juan Ramón Jiménez, Huelva; Gonzalo Gómez Gómez, MD, Principal Investigator — Hospital Universitario 12 de Octubre, Madrid; Daniel Carpio López, MD, Principal Investigator — Hospital de Montecelo, Pontevedra; Xavier Cortés Rizo, MD, Principal Investigator — Hospital de Sagunto, Valencia; Torsten Kucharzik, Professor, Principal Investigator — Klinikum Lüneburg; Andreas Sturm, Professor, Principal Investigator — Krakenhaus Walfriede, Berlin; Antonio López Sanromán, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Joaquín Hinojosa de Val, MD, Principal Investigator — Hospital de Manises, Valencia; Xavier González Argenté, MD, Principal Investigator — Son Espases, Palma de Mallorca; Maria Nachury, MD, Principal Investigator — CHRU de Lille; Frank Zerbib, MD, Principal Investigator — University Hospital, Bordeaux; Stéphanie Viennot, MD, Principal Investigator — University Hospital, Caen; Jean-Louis Dupas, MD, Principal Investigator — Centre Hospitalier Universitaire, Amiens; Jean-Charles Grimaud, MD, Principal Investigator — CHU de Marseille; Xavier Hebuterne, Professor, Principal Investigator — Centre Hospitalier Universitaire de Nice; Matthieu Allez, Professor, Principal Investigator — Hôpital Saint Louis Paris; Yoram Bouhnik, MD, Principal Investigator — Hôpital Beaujon, Clichy; Matti Waterman, MD, Principal Investigator — Rambam MC, Haifa; Shomron Ben-Horin, MD, Principal Investigator — Sheba MC, Tel Hashomer; Sigal Fishman, MD, Principal Investigator — Tel Aviv Sourasky MC, Tel Aviv; Eran Goldin, Professor, Principal Investigator — Sharee Zedek MC, Jerusalem; Irit Avni-Biron, MD, Principal Investigator — Rabin MC, Petah Tikva; Herbert Tilg, Professor, Principal Investigator — Univ.-Klinik Innsbruck; Lennard Gilissen, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Carlos Pastor, MD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz; Wolfgang Kruis, Professor, Principal Investigator — Evangelisches Krankenhaus Kalk, Köln
Locations (52):
- Austria (3):
  - Univ.-Klinik Innsbruck, Innsbruck
  - Krankenhaus, Saint Veit/Glan
  - Medizinische Universität, Vienna
- Belgium (4):
  - Hospital Oost-Limburg, Genk
  - Gent University Hospital, Ghent
  - Leuven University Hospital, Leuven
  - Hospital Hartziekenhuis, Roeselare
- France (8):
  - CHU d'Amiens, Amiens
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - Hôpital Beaujon, Clichy
  - CHRU de Lille, Lille
  - CHU de Marseille, Marseille
  - CHU de Nice, Nice
  - Hôpital Saint-Louis, Paris
- Germany (6):
  - Charite, Berlin
  - Krakenhaus Walfriede, Berlin
  - Klinikum Braunscheweig, Braunschweig
  - Evangelisches Krankenhaus Kalk, Cologne
  - Klinikum Frankfurt, Frankfurt am Main
  - Klinikum Lüneburg, Lüneburg
- Israel (5):
  - Rambam MC, Haifa
  - Sharee Zedek MC, Jerusalem
  - Rabin MC, Petah Tikva
  - Tel Aviv Sourasky MC, Tel Aviv
  - Sheba MC, Tel Litwinsky
- Italy (7):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Instituto Clinico Humanitas IRCCS, Milan
  - Seconda Università degli Studi di Napoli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera San Camillo-Forlanini, Rome
  - Università Cattolica del Sacro Cuore, Rome
- Netherlands (4):
  - AMC, Amsterdam
  - VUMC, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - UMCU, Utrecht
- Spain (15):
  - Hospital de Manises, Manises, Valencia
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Juan Ramon Jimenez, Huelva
  - Hospital Ramón y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Son Espases, Palma de Mallorca
  - Hospital de Montecelo, Pontevedra
  - Hospital Virgen del Rocio, Seville
  - Hospital de Sagunto, Valencia
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Derived] Garcia-Olmo D, Gilaberte I, Binek M, D Hoore AJL, Lindner D, Selvaggi F, Spinelli A, Panes J. Follow-up Study to Evaluate the Long-term Safety and Efficacy of Darvadstrocel (Mesenchymal Stem Cell Treatment) in Patients With Perianal Fistulizing Crohn's Disease: ADMIRE-CD Phase 3 Randomized Controlled Trial. Dis Colon Rectum. 2022 May 1;65(5):713-720. doi: 10.1097/DCR.0000000000002325. PMID 34890373
- [Derived] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Derived] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896